CLINICAL TRIAL: NCT04406493
Title: Monitoring of Lung Fluid Status of Hospitalized COVID-19 Patients by Lung Impedance Technique
Brief Title: Monitoring COVID-19 Patients' Lung Fluid Using Impedance Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0059-20-HYMC
Record Dates: First submitted 2020-05-23; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: ARDS; COVID

STUDY DESIGN:
Intervention Model Description: COVID 19 patients are admitted to Infectious Diseases Unit, will undergo examination using lung impedance device. The first value that has been measured will be set as BASAL.
  During the hospitalization each patient will undergo this examination twice a day until discharged.
  Changes in impedance values during admission will be evaluated as POSITIVE AND NEGATIVE PREDICTIVE values for clinical deterioration and improvement of COVID 19 patients and as a factor which predicts mechanical ventilation The time between lung impedance started to decrease (expression of the lung fluids accumulation) and the need in mechanical ventilation will be measured.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID 19 patients (Experimental): COVID 19 patients are admitted to the Infectious Diseases Unit, will undergo examination using a lung impedance device. The first value that has been measured will be set as BASAL.
  During the hospitalization each patient will undergo this examination twice a day until discharged.
  Changes in impedance values during admission will be evaluated as POSITIVE AND NEGATIVE PREDICTIVE values for clinical deterioration and improvement of COVID 19 patients and as a factor which predicts mechanical ventilation The time between lung impedance started to decrease (expression of the lung fluids accumulation) and the need for mechanical ventilation will be measured.
  Interventions: Diagnostic Test: Lung impedance technique

INTERVENTIONS:
Diagnostic Test: Lung impedance technique — COVID 19 patients are admitted to the Infectious Diseases Unit; they will undergo examination using a lung impedance device. The first value that has been measured will be set as BASAL.
  During the hospitalization, each patient will undergo this examination twice a day until discharge.
  Changes in impedance values during admission will be evaluated as POSITIVE AND NEGATIVE PREDICTIVE values for clinical deterioration and improvement of COVID 19 patients and as a factor which predicts mechanical ventilation.
  The time between lung impedance started to decrease (expression of the lung fluids accumulation), and the need for mechanical ventilation will be measured.

SUMMARY:
COVID 19 is a novel and severe disease. One of the problems is that the virus disturbs the lungs and cause water accumulation in lungs alveolus (ARDS).

Today, a chest X-ray is the only practical way to check the degree of lung accumulation. However, X-Ray has many limitations and disadvantages.

Lung impedance technology allows simple lung fluid monitoring, and found to be effective in HF patients who suffer from a similar problem.

The study's aim is to establish a correlation between lung fluid assessed by impedance technique and x-ray examinations. To find a correlation between lung fluid assessment by impedance and clinical parameters of COVID 19 patients.

DETAILED DESCRIPTION:
COVID 19 is a novel and severe disease. One of the problems is that the virus disturbs the lungs and cause water accumulation in lungs alveolus (ARDS). Water accumulation in pulmonary alveoli leads to fast deterioration and, eventually death. It is important to note that at an early stage of the disease, when the patient feels relatively good, fluid progressively accumulates into the lung.

Today chest X-ray is the only practical way to check the degree of lung accumulation. Chest X ray is a cumbersome method and has a rotational burden. One of the disadvantages of the x-ray is that interpretation of x-ray results are operator dependent. Another disadvantage is the daily monitoring of lung fluids, which is expensive.

Lung impedance technology allows simple lung fluid monitoring, and found to be effective in HF patients who suffers from the same problem, fluid accumulation in lungs. Lung fluid monitoring using lung impedance device may assist physicians to reveal fluid accumulation in lungs, and give better understanding of the severity of the situation. Moreover, better impedance values indicate improvement in patient's condition and also effectiveness of the treatment.

The aim of the study is to prove the correlation between lung fluid assessed by impedance technique and x-ray examinations. To find correlation between lung fluid assessment by impedance and clinical parameters of COVID 19 patients.

In a case that this correlation would be found high, then it will be possible to establish monitoring of lung fluid status of COVID 19 patients using lung impedance device, as a simple and reliable way to determine degree of patient's deterioration as it was proved for HF patients.

The main question, is if a changes in lung fluid status assessed by impedance technique may indicate the need in artificial respiration before there is a drastic Deterioration in patient's condition.

COVID 19 patients are admitted to Infectious Diseases Unit, will undergo examination using lung impedance device. The first value that has been measured will be set as BASAL.

During hospitalization, each patient will undergo this examination twice a day until discharged.

Changes in impedance values during admission will be evaluated as POSITIVE AND NEGATIVE PREDICTIVE values for clinical deterioration and improvement of COVID 19 patients and as a factor that predicts mechanical ventilation.

The time between lung impedance started to decrease (expression of the lung fluids accumulation), and the need in mechanical ventilation will be measured.

In a case that lung impedance would be found as a useful predictor of clinical condition in COVID 19 patients, the application for second stage of the study will be submitted to Helsinki Committee.

On the second stage of the study is planning to use lung impedance values as guide for the decision about beginning mechanical ventilation of COVID 19 patients before critical deterioration.

Each patient which is hospitalized in Infectious Diseases Unit of Hillel Yaffe Medical Center suitable for study.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 patient admitted to the infectious unit

Exclusion Criteria:

* patients who do not agree to sign informed consent, or participating in other studies.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-04-28 (Estimated); Study Completion 2021-04-28 (Estimated)

PRIMARY OUTCOMES:
Correlation between impudence deterioration to clinical conditions and hospitalization period | Estimated a month, but could be prolonged through the study completion (one year)
  the changes in lung fluid status assessed by impedance technique will be compared to the patient's clinical conditions and the patient's length of stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe MC,, Hadera, Israel

IPD SHARING:
Plan to Share IPD: Undecided